CLINICAL TRIAL: NCT04166955
Title: WhatsApp-Based Intervention for Promoting Physical Activity Among Female College Students, Saudi Arabia: A Randomized Controlled Trial
Brief Title: What'Sapp Based Intervention for Promoting Physical Activity Among Female College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Amal Alshahrani, Principal investigator, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H06B091
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Intervention) (Experimental): Participants will be provided with weekly messages including information for promoting physical activity.
  Interventions: Behavioral: Promoting Physical Activity through mobile application
- (Control) (No Intervention): Participants will be evaluated without providing any intervention.

INTERVENTIONS:
Behavioral: Promoting Physical Activity through mobile application — Students will be randomly assigned to either the intervention or the control group. WhatsApp groups will be formed within each study group. The control participants will have the WhatsApp group only for communications. And they will keep their usual activity for 10 weeks. The intervention participants will have the intervention WhatsApp group which will be for communication and providing the intervention materials. The intervention group will receive a brief (15-minute) orientation on exercise, and benefits of keeping a healthy life pattern. They will receive 3-4 health-promotional (Physical activity) messages per week via WhatsApp for 10 weeks; group interaction is optional without adding more messages aiming to promote physical activities from any participants.
  Arms: (Intervention)

SUMMARY:
The purpose of this research will be to determine the efficacy and applicability of using WhatsApp-based intervention for physical activity promotion in female college students.

DETAILED DESCRIPTION:
In the recent past, adoption of social media as a way of daily communication has been on the rise. For instance, according to Ventiola the healthcare sector has many social media tools including networking platforms, Wikis, blogs, media sharing sites, and virtual reality and gaming sites . These tools are necessary for improving the practice of healthcare workforce by promoting real time interaction, patient education, as well as public health education. However, the social media tools also present potential risk to patients including breach of patient information safety and also extension of professional boundaries to personal levels . However, as a revolutionary communication tool, social media has enhanced patient-practitioner relationship by ensuring that the two connect even outside the healthcare environment. Therefore, the application of social media in healthcare management and dissemination of services is not by accident, but rather, a timely invention that will see the improvement of health standards globally if well implemented.

It is essential to first understand the meaning of social media before any of its application in promoting client-practitioner relationship is discussed. It is even more necessary when the issue is related to healthcare management since the dissemination of healthcare services is a critical affair. According to Kaplan and Michael social media is "a group of Internet-based applications that build on the ideological and technological foundations of Web 2.0 which allows the creation and exchange of User Generated Content." However, the new perspective should not make researchers drool on the fact that social media is Web 2.0 based; rather, the meaning of social media must be expanded to include both online and offline social activities. Thus, social media can be considered as a versatile communication tool that allows for interactive communication based on personal experiences that aim at influencing the actions of each other .

Based on that context, it is imperative to note that the use of social media in healthcare management is not so common due to myriad factors that cannot be expressly identified. However, it is understandable that social media and its level of sophistication today, is ripe for social support in any human engagement. Thus, due to its versatility, reach and functionality, social media now qualifies as the most promising online support tool with minimum resource uptake. Most importantly, the recent studies indicate that social media has succeeded elsewhere in helping certain individuals meet their social and health goals thus making the subject worth a more profiled review. Physical activity is now a well-established element of the public health agenda. today's university students are our future social opinion leaders and policy makers and as such, their habits, beliefs and attitudes will be influential in shaping community norms and values. In addition, as a group, they are spending considerable time in a setting that promotes sedentary behavior (particularly computer and Internet use) and are largely being educated for sedentary occupations .

Adherence to physical activity (PA) leads to improvements in physical function and quality of life . The adherence is one of the most important factors in order to get the desired benefits of PA. The role of the PA has been well- discussed in several studies and found to aid prevention of many health disorders, such as cardiovascular diseases and obesity . Regular exercise, in particular, helps protect against debilitating and costly chronic conditions as well and to achieve the optimum level of quality of life . Adherence to PA must be improved in order to improve health prospects. The adherence to the PA has been found to be extremely low in the Saudi population, particularly among young females . This poor adherence could be attributable to lack of knowledge about the benefits of exercise or even many related social and personal factors as well as cultural factors . The dangers of physical inactivity have been outlined in many studies as it is one of the most important public health problems of the 21st century . For example, physically inactive middle-aged women (performed less than 1 hour of exercise per week) experienced 52% increased all-cause mortality, a doubling of cardiovascular related mortality and 29% increased cancer-related mortality compared with the physically active women . Motivation for PA could be defined as the intrinsic and extrinsic factors that stimulate desire and energy in people to be continually interested and committed to the initiation and the maintenance of a PA program or any type of exercise (10). Intrinsically motivated behaviors are those performed for satisfaction one gains from engaging in the activity itself. By contrast, extrinsically motivated behaviors are those performed in order to get rewards or results that are separate from the behavior itself . There are many different ways that have been used to increase the adherence level to the PA and the home exercise programs are an effective motivational way . Previous studies reported positive effect of using electronic media and mobile phone applications to enhance motivation in improving adherence among participants . Fukuoka et al. investigated the use of mobile phone based intervention to improve physical activity in sedentary women. They concluded that the mobile phone based intervention seems to motivate inactive women to improve their physical activity. Another study reported significant effects of Internet and mobile phone based motivation to improve the level of physical activity in healthy adults . In addition, Turner-McGreevy et al. reported some potential benefits of mobile phone monitoring methods during weight reduction intervention in overweight adults . The present study aimed primarily to evaluate the efficacy of using social media "WhatsApp application" as a motivational stimulus in improving Physical Activity levels among Saudi female college students in Abha city.

ELIGIBILITY:
Inclusion Criteria:

* Being a female student studying at King Khaled University.
* Age range from 18 Years to 28 Years.
* owns smartphone with internet access and WhatsApp application.
* Willing to complete all study requirement.

Exclusion Criteria:

* Physical disability that precludes physical activity.
* Morbidly obese (Body Mass Index >45 kg/m2)
* Physician recommendation not to exercise.
* pregnant female

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Self-reported physical activity | Time Frame: Baseline to 10 weeks follow-up
  Change between baseline and follow-up for physical activity . Measurement tool = Global Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- king khaled University, Abhā, Asir Providences, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventola CL. Social media and health care professionals: benefits, risks, and best practices. P T. 2014 Jul;39(7):491-520. PMID 25083128
- [Background] Nelson S, Heyder AM, Stone J, Bergeron MG, Daugherty S, Peterson G, Fotheringham N, Welch W, Milwee S, Root R. A randomized controlled trial of filgrastim for the treatment of hospitalized patients with multilobar pneumonia. J Infect Dis. 2000 Sep;182(3):970-3. doi: 10.1086/315775. Epub 2000 Aug 17. PMID 10950800
- [Background] Martinsen EW. Physical activity in the prevention and treatment of anxiety and depression. Nord J Psychiatry. 2008;62 Suppl 47:25-9. doi: 10.1080/08039480802315640. PMID 18752115
- [Background] Hu G, Barengo NC, Tuomilehto J, Lakka TA, Nissinen A, Jousilahti P. Relationship of physical activity and body mass index to the risk of hypertension: a prospective study in Finland. Hypertension. 2004 Jan;43(1):25-30. doi: 10.1161/01.HYP.0000107400.72456.19. Epub 2003 Dec 1. PMID 14656958
- [Background] Al-Nozha MM, Al-Hazzaa HM, Arafah MR, Al-Khadra A, Al-Mazrou YY, Al-Maatouq MA, Khan NB, Al-Marzouki K, Al-Harthi SS, Abdullah M, Al-Shahid MS. Prevalence of physical activity and inactivity among Saudis aged 30-70 years. A population-based cross-sectional study. Saudi Med J. 2007 Apr;28(4):559-68. PMID 17457478
- [Background] Al-Eisa ES, Al-Sobayel HI. Physical Activity and Health Beliefs among Saudi Women. J Nutr Metab. 2012;2012:642187. doi: 10.1155/2012/642187. Epub 2012 Feb 22. PMID 22523673
- [Background] Turner-McGrievy GM, Beets MW, Moore JB, Kaczynski AT, Barr-Anderson DJ, Tate DF. Comparison of traditional versus mobile app self-monitoring of physical activity and dietary intake among overweight adults participating in an mHealth weight loss program. J Am Med Inform Assoc. 2013 May 1;20(3):513-8. doi: 10.1136/amiajnl-2012-001510. Epub 2013 Feb 21. PMID 23429637
- [Background] Alahmed Z, Lobelo F. Physical activity promotion in Saudi Arabia: A critical role for clinicians and the health care system. J Epidemiol Glob Health. 2018 Mar;7 Suppl 1(Suppl 1):S7-S15. doi: 10.1016/j.jegh.2017.10.005. Epub 2017 Oct 24. PMID 29801594
- [Background] Zhang J, Brackbill D, Yang S, Centola D. Efficacy and causal mechanism of an online social media intervention to increase physical activity: Results of a randomized controlled trial. Prev Med Rep. 2015 Aug 13;2:651-7. doi: 10.1016/j.pmedr.2015.08.005. eCollection 2015. PMID 26844132
- [Background] Al-Eisa E, Al-Rushud A, Alghadir A, Anwer S, Al-Harbi B, Al-Sughaier N, Al-Yoseef N, Al-Otaibi R, Al-Muhaysin HA. Effect of Motivation by "Instagram" on Adherence to Physical Activity among Female College Students. Biomed Res Int. 2016;2016:1546013. doi: 10.1155/2016/1546013. Epub 2016 Feb 29. PMID 27034927